CLINICAL TRIAL: NCT06480929
Title: Left Ventricular Thrombus Routine Screening With Contrast Echocardiography in Patients With Anterior ST-elevation Myocardial Infarction: is it Worth it?
Brief Title: LV Thrombus Screening in Anterior STEMI: Worth it?
Acronym: LVT-CE-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Tondela-Viseu (Other)
Responsible Party: Principal Investigator, Joana Maria Laranjeira Correia, Dr., Centro Hospitalar Tondela-Viseu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHTondelaViseu
Record Dates: First submitted 2024-06-21; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Thrombus of Left Ventricle; Anterior Wall Myocardial Infarction; ST Elevation Myocardial Infarction; Echocardiography
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Active Comparator): The study group included all patients admitted on odd numbered days of the month that performed a contrast TTE,
  Interventions: Other: Contrast TTE procedure, the SonoVue ultrasound agent
- control group (No Intervention): The control group included patients admitted on even numbered days and were submitted to a conventional

INTERVENTIONS:
Other: Contrast TTE procedure, the SonoVue ultrasound agent — The intervention involved using contrast-enhanced transthoracic echocardiography (TTE) to improve the detection of left ventricular thrombus in patients with anterior ST-elevation myocardial infarction (STEMI).
  Arms: study group

SUMMARY:
Left ventricular (LV) thrombus is more common in patients with anterior ST-elevation myocardial infarction (STEMI) compared to other types of acute myocardial infarction (AMI) and is linked to worse outcomes. Diagnosing LV thrombus remains challenging. Contrast echocardiography (TTE) has potential to improve diagnostic accuracy, affecting treatment strategies involving antithrombotic/anticoagulation therapy.

This study aimed to evaluate the effectiveness of contrast TTE as a routine screening method for detecting LV thrombus in the acute phase of anterior STEMI.

DETAILED DESCRIPTION:
The advent of primary percutaneous coronary intervention (PCI) has significantly lowered mortality rates associated with acute myocardial infarction (AMI). Despite these advancements, post-infarction complications, including left ventricular (LV) thrombus, continue to negatively impact prognosis. The incidence of LV thrombus has decreased due to improved reperfusion techniques and antithrombotic therapies; however, it remains a significant risk factor for embolic events, with up to a 10% risk of stroke within a year despite anticoagulation therapy. The formation of thrombus post-AMI, particularly in anterior ST-elevation myocardial infarction (STEMI), is driven by endothelial injury, blood stasis due to LV dysfunction, and hypercoagulability from inflammation.

Anterior STEMI, usually caused by occlusion of the left anterior descending artery, often leads to LV apical akinesia and subsequent thrombus formation within 24 hours to two weeks post-AMI. Guidelines recommend routine transthoracic echocardiography (TTE) post-PCI to evaluate LV function and detect early post-infarction mechanical complications and LV thrombus. However, conventional TTE can be limited by operator skill and may miss thrombi, especially in cases with suboptimal images or small/mural thrombi. Advances in ultrasound technology, including contrast agents, have improved diagnostic accuracy for LV thrombus by enhancing LV opacification and endocardial border delineation, thus identifying the characteristic "filling defect" of intracardiac thrombus.

This study aimed to assess the effectiveness of contrast-enhanced TTE as a routine screening method for detecting LV thrombus in the acute phase of anterior STEMI.

A prospective, single-center, randomized controlled trial was conducted with patients admitted for anterior STEMI at Centro Hospitalar de Tondela-Viseu from November 2021 to January 2023. Patients were randomly assigned to a study group (undergoing contrast TTE) or a control group (undergoing conventional TTE). Exclusion criteria included patients under 18, those without echocardiographic or coronary angiographic evaluation, those with cardiogenic shock, known thrombus, or allergic reactions to contrast agents. Contrast TTE utilized the SonoVue ultrasound agent and GE i9 echocardiograph, performed by specialized cardiologists. Data collected included demographic, clinical, and procedural information, with statistical analysis comparing the characteristics and outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Admitted due to anterior ST-elevation myocardial infarction

Exclusion Criteria:

* Under 18 years old
* Did not undergo echocardiographic or coronary angiographic evaluation
* Cardiogenic shock
* Previously known thrombus
* Previously known allergic contrast reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
left ventricular thrombus | 7 days (time of echoTT)
  Presence or absence of left ventricular thrombus detected via transthoracic echocardiography with or without contrast agent during hospital admission for acute anterior ST-elevation myocardial infarction (STEMI)

SECONDARY OUTCOMES:
anterior/apical aneurysm | 7 days (time of echoTT)
  Presence or absence of anterior/apical aneurysm confirmed by echocardiography with or without contrast agent during hospital admission for acute anterior ST-elevation myocardial infarction (STEMI) and at follow-up visits post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Joana ML Correia, Principal Investigator — 219827419
Locations (1):
- Centro Hospitalar Tondela Viseu, Viseu, Visey, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected during this study will be handled with confidentiality and privacy protection measures in place. Due to the sensitive nature of health information, access to IPD will be restricted to authorized personnel only, in accordance with ethical guidelines and regulatory requirements. Researchers interested in accessing the anonymized data for further analysis or collaboration may contact the principal investigator directly after publication, following established data sharing protocols and agreements.

REFERENCES:
- [Derived] Correia JL, Ferreira GRM, Fiuza JG, Almeida MD, Coelho J, Correia E, Correia JM, Moreira D, Craveiro N, Goncalves ML, Neto VD. Left ventricular thrombus routine screening with contrast echocardiography in patients with anterior ST-elevation myocardial infarction: is it worth it? J Cardiovasc Imaging. 2024 Aug 5;32(1):21. doi: 10.1186/s44348-024-00027-0. PMID 39103940